CLINICAL TRIAL: NCT02409823
Title: Clinical Registry of Patients Under Treatment With Atypical Antipsychotics
Status: Completed | Type: Observational
Sponsor: Pontifical Catholic University of Argentina (Other)
Responsible Party: Principal Investigator, Santiago Perez Lloret, MD PhD CPI, Pontifical Catholic University of Argentina
Other Study IDs: 1209-Re03-Reg
Record Dates: First submitted 2015-04-01; First posted 2015-04-07 (Estimated); Last update posted 2015-10-20 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia; Major Depressive Disorder; Bipolar Depressive Disorder; Parkinson's Disease With Hallucinations
Keywords: adverse drug reactions; adherence to treatment; quality of life; clinical status
MeSH Terms: conditions — Schizophrenia; Depressive Disorder, Major; Drug-Related Side Effects and Adverse Reactions; Treatment Adherence and Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients on atypical antipsychotics
  Interventions: Drug: Atypical Antipsychotics

INTERVENTIONS:
Drug: Atypical Antipsychotics — any atypical antipsychotic

SUMMARY:
Antipsychotic drugs are characterized by blocking dopaminergic D2 receptors. They have been found to be effective and safe for the treatment of schizophrenia, bipolar disorders, depressive episodes associated with bipolar disorder, or psychotic symptoms in the context of Parkinson's disease. Atypical antipsychotics have lower blocking potency on D2 receptors, at the time that interact with serotoninergic, adrenergic and histaminergic receptors, among others. Quetiapine extended-release has the same clinical efficacy as the immediate-release formulation, but reduces the amount of daily doses, possibly contributing to increased treatment adherence.

The purpose of this registry is to explore adherence to treatment, the occurrence of adverse drug reactions and the clinical outcomes in a sample of patients under treatment with atypical antipsychotics in several Central American countries. For this study, clinical data will be extracted from the medical records of 1000 patients with schizophrenia, depressive disorders or Parkinson's Disease with hallucinations. Occurrence of adverse drug reactions, namely weight gain, somnolence, extrapyramidal reactions and symptoms of orthostatic hypotension; adherence to treatment; and changes in quality of life and clinical status will be assessed during the first 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years-old
* have a diagnosis of schizophrenia, major depressive disorder, bipolar depressive disorder, parkinson's disease with hallucination
* such patients should receive antipsychotics as their usual treatment
* they should give informed consent before participating

Exclusion Criteria:

* no treatment with atypical antypsichotics
* other diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients under atypical antipsychotic therapy
Sampling Method: Non-Probability Sample
Enrollment: 665 (Actual)
Dates: Start 2015-02; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of Adverse Drug Reactions | 8 weeks
Adherence to treatment | 8 weeks

SECONDARY OUTCOMES:
Quality of Life | 8 weeks
Clinical status (CGI score) | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Santiago Perez Lloret, MD PhD CPI, Principal Investigator — Pontifical Catholic University of Argentina

REFERENCES:
- [Derived] Rey MV, Molina L, Recinos B, Paz B, Rovelo M, Rodriguez Elias FE, Calderon J, Arellano A, Perez-Lloret S; CA-APD Study Team. Movement Disorders After Exposure to Antipsychotic Drugs in Patients With Depressive Disorders. Clin Neuropharmacol. 2018 Sep/Oct;41(5):177-180. doi: 10.1097/WNF.0000000000000300. PMID 30234617
- [Derived] Molina L, Recinos B, Paz B, Rovelo M, Elias Rodriguez FE, Calderon J, Arellano A, Pomata S, Rey MV, Perez-Lloret S. Factors Related to Early Clinical Effects of Quetiapine Extended-Release: A Multinational, Prospective, Observational Study. Clin Drug Investig. 2016 Jun;36(6):491-7. doi: 10.1007/s40261-016-0395-x. PMID 27021967